CLINICAL TRIAL: NCT01339936
Title: Evaluation of the Effect of Repeated Usage on the Tear Film Characteristics of an Investigational Eye Drop in Dry Eye Sufferers
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Optometric Technology Group Ltd (Other)
Collaborators: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: AG9965-005 ID 10-12
Record Dates: First submitted 2011-04-19; First posted 2011-04-21 (Estimated); Results first posted 2013-11-28 (Estimated); Last update posted 2013-11-28 (Estimated); Status verified 2013-09

CONDITIONS: Dry Eye Syndrome
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Investigational eye drop (Experimental): Formulation 1: Carboxymethylcellulose sodium, glycerin and polysorbate 80 based eye drops formulated for the relief of ocular surface irritation and symptoms of dryness
  Interventions: Device: Carboxymethylcellulose sodium, glycerin and polysorbate 80

INTERVENTIONS:
Device: Carboxymethylcellulose sodium, glycerin and polysorbate 80 — 1 drop in each eye three times a day for a period of 30 (± 4) days

SUMMARY:
The main objectives of the investigation will be to assess the effect of the repeated usage of an investigational eye drop on the tear film characteristics of dry eye sufferers and demonstrate the benefit of this eye drops for dry eye sufferers.

ELIGIBILITY:
Inclusion Criteria:

* Mild or greater dry eye symptoms.
* Evidence of evaporative dry eye

Exclusion Criteria:

* Known allergy or sensitivity to the study product(s) or its components
* Current contact lens wearer
* Systemic or ocular allergies
* Use of systemic medication which might have ocular side effects.
* Any ocular infection.
* Use of ocular medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-03; Primary Completion 2011-08 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- OTG Research & Consultancy, London, England, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The subjects were selected from the existing clinical population of Optometric Technology Group Ltd (OTG Research & Consultancy). The subjects, fulfilling the criteria for inclusion were invited in a random fashion to participate in the study until the test population was achieved.
Period: Overall Study
Arm/Group | Investigational Eye Drop
Started | 38 (plus 2 screen failures)
Completed | 36 (plus 1 excluded from analysis set)
Not Completed | 2

BASELINE CHARACTERISTICS:
Population: The analysis was per protocol hence on 35 participants
Arm/Group | Investigational Eye Drop
Number analyzed (Participants) | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 28
  >=65 years | 6
Age Continuous [Mean (Standard Deviation); unit: years] | 49 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 8
Region of Enrollment [Number; unit: participants]
  United Kingdom | 35

OUTCOME MEASURES:

1. Primary Outcome: Tear Film Evaporation Rate
Description: The rate of evaporation of the tears from the ocular surface was measured. To do so the participant was required to wear a sealed goggle over the eye, which served to isolate the air surrounding the ocular surface. The temperature and humidity were measured within the sealed goggle during closed eye and open eye situations. The evaporation from the ocular surface was calculated by taking the difference between the evaporation rate of the skin taken during the closed eye measurement and the evaporation rate taken during the open eye measurement. The rate of evaporation was measured in 10^-7 g/cm^2 /s and recorded for relative humidity of 25% to 35%.
Time Frame: after 30 days of eyedrop usage
Population: The analysis was carried out on subjects having completed the study according to the protocol e.g. 35
Measure: Mean (Standard Deviation); unit: 10^-7g/cm^2/sec
Arm/Group | Investigational Eye Drop
Number analyzed (Participants) | 35
10^-7g/cm^2/sec | 26.0 (11.2)

2. Secondary Outcome: Tear Break Up Time
Description: The tear film break-up-time (BUT) is the time elapsed between eye opening after a blink, and the appearance of the first dark spot within the tear film when observed with a wide diffuse light source of the Tearscope. This measurement is indicative of the tear film stability. Three independent measurements were recorded in each case and the median value over the three measurements calculated. The latter value constituted the secondary endpoint used in the analysis.
Time Frame: after 30 days of eyedrop usage
Population: The analysis was carried out on subjects having completed the study according to the protocol e.g. 35
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Investigational Eye Drop
Number analyzed (Participants) | 35
seconds | 5.8 (4.3)

3. Secondary Outcome: Ocular Surface Disease Index Score
Description: The OSDI is a 12-item patient-reported outcomes questionnaire designed to assess the range of ocular surface symptoms, their severity, and their impact on the patient's ability to function.
  The OSDI items are scored on a 0 to 4 Likert-type scale, where 0 = None of the time, 1 = Some of the time, 2 = Half of the time, 3 = Most of the time, and 4 = All of the time. Using individual item responses, an overall OSDI score is calculated. The overall OSDI score ranges from 0 to 100, where a score of 100 corresponds to complete disability while a score of 0 corresponds to no disability.
Time Frame: after 30 days of eye drop usage
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Investigational Eye Drop
Number analyzed (Participants) | 35
points | 26.8 (23.0)

ADVERSE EVENTS:
Arm/Group | Investigational Eye Drop
Serious Adverse Events (participants affected / at risk) | 0/36
Other Adverse Events (participants affected / at risk) | 3/36
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Investigational Eye Drop (N=36)
Stye (Eye disorders) | 1 (1)
Allergic response (Skin and subcutaneous tissue disorders) | 1 (1)
Bunion surgery (Surgical and medical procedures) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication policy

The investigation data is wholly owned by the Sponsor. The results of the investigation may not be used in publications or presentations without the written permission of the Sponsor.